CLINICAL TRIAL: NCT05952856
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of MK-0616 in Adults With Hypercholesterolemia
Brief Title: A Study of Enlicitide Decanoate (MK-0616 Oral PCSK9 Inhibitor) in Adults With Hypercholesterolemia (MK-0616-013) CORALreef Lipids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0616-013; MK-0616-013 (Other: MSD); 2022-502777-42-00 (Registry Identifier: EU CT); U1111-1285-4164 (Registry Identifier: UTN); jRCT2031230320 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2023-07-10; First posted 2023-07-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hypercholesterolemia; Familial Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — MK-0616

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enlicitide Decanoate (Experimental): Participants will receive 20 mg of enlicitide decanoate orally once daily (QD) for up to 52 weeks.
  Interventions: Drug: Enlicitide Decanoate
- Placebo (Placebo Comparator): Participants will receive enlicitide decanoate-matching placebo orally QD for up to 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enlicitide Decanoate — Oral tablet
  Other Names: MK-0616
  Arms: Enlicitide Decanoate
Drug: Placebo — Oral tablet
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate the efficacy, safety, and tolerability of enlicitide decanoate in adult participants with hypercholesterolemia. The primary hypothesis is that enlicitide decanoate is superior to placebo on mean percent change from baseline in low-density lipoprotein cholesterol (LDL-C) at Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Has a history of a major atherosclerotic cardiovascular disease (ASCVD) event and LDL-C ≥55 mg/dL OR, if no history of a major ASCVD event, has intermediate to high risk for development of a first major ASCVD event and LDL-C ≥70 mg/dL.
* Is treated with a moderate- or high-intensity statin OR is treated with low-intensity statin with documentation of intolerance to a moderate or high-intensity statin OR is not receiving statins with documentation of statin intolerance
* If on any lipid-lowering therapies (LLTs), should be on a stable dose with no planned medication change.

Exclusion Criteria:

* Has a history of homozygous familial hypercholesterolemia (FH) based on genetic or clinical criteria, compound heterozygous FH, or double heterozygous FH
* Has a history of heart failure or heart failure hospitalization within 3 months before first study visit
* Is undergoing or previously underwent an LDL-C apheresis program within 3 months before first study visit or plans to initiate an LDL-C apheresis program
* Was previously treated/is being treated with certain other cholesterol lowering medications, including protein convertase subtilisin/kexin type 9 (PCSK9) inhibitors without adequate washout

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2912 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Mean percent change from baseline in low-density lipoprotein cholesterol (LDL-C) at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess mean percent change in LDL-C.
Number of participants with one or more adverse events (AEs) | Up to ~60 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study drug due to an AE | Up to ~52 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Mean percent change from baseline in LDL-C at Week 52 | Baseline and Week 52
  Blood samples will be collected at baseline and at Week 52 to assess mean percent change in LDL-C.
Mean percent change from baseline in non-high-density lipoprotein cholesterol (non-HDL-C) at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess mean percent change in non-HDL-C.
Mean percent change from baseline in apolipoprotein B (ApoB) at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess mean percent change in ApoB.
Percent change from baseline in lipoprotein(a) (Lp[a]) at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess percent change in Lp(a).
Percentage of participants with LDL-C <70 mg/dL and ≥50% reduction from baseline at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess the percentage of participants who have LDL-C <70 mg/dL and ≥50% reduction from baseline.
Percentage of participants with LDL-C <55 mg/dL and ≥50% reduction from baseline at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess the percentage of participants who have LDL-C <55 mg/dL and ≥50% reduction from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (168):
- United States (49):
  - Alliance for Multispecialty Research, LLC ( Site 0093), Daphne, Alabama
  - G&L Research ( Site 0043), Foley, Alabama
  - Synexus Clinical Research US, Inc.-Synexus Clinical Research US, Inc - Central Phoenix ( Site 0084), Phoenix, Arizona
  - National Heart Institute-Research ( Site 0087), Beverly Hills, California
  - Clinical Trials Research ( Site 0115), Sacramento, California
  - Velocity Clinical Research, Banning ( Site 0017), San Bernardino, California
  - Emerson Clinical Research Institute ( Site 0118), Washington D.C., District of Columbia
  - Excel Medical Clinical Trials ( Site 0053), Boca Raton, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0088), Coral Gables, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0094), Fort Myers, Florida
  - Velocity Clinical Research, Hallandale Beach ( Site 0018), Hallandale, Florida
  - Jacksonville Center for Clinical Research ( Site 0049), Jacksonville, Florida
  - South Broward Research ( Site 0051), Miramar, Florida
  - Clinical Research Trials of Florida ( Site 0063), Tampa, Florida
  - East Coast Institute for Research, LLC ( Site 0033), Macon, Georgia
  - Healthcare Research Network - Chicago ( Site 0052), Flossmoor, Illinois
  - Synexus Clinical Research US, Inc. ( Site 0109), Evansville, Indiana
  - Midwest Institute For Clinical Research ( Site 0059), Indianapolis, Indiana
  - Alliance for Multispecialty Research, LLC ( Site 0028), Lexington, Kentucky
  - L-MARC Research Center ( Site 0001), Louisville, Kentucky
  - Velocity Clinical Research, Covington ( Site 0068), Covington, Louisiana
  - Velocity Clinical Research Rockville ( Site 0082), Rockville, Maryland
  - Velocity Clinical Research, Gulfport ( Site 0039), Gulfport, Mississippi
  - Healthcare Research Network - St. Louis ( Site 0054), Hazelwood, Missouri
  - Jubilee Clinical Research ( Site 0106), Las Vegas, Nevada
  - AB Clinical Trials ( Site 0070), Las Vegas, Nevada
  - New Mexico Clinical Research & Osteoporosis Center ( Site 0005), Albuquerque, New Mexico
  - Velocity Clinical Research, Syracuse ( Site 0021), East Syracuse, New York
  - Icahn School of Medicine at Mount Sinai-Cardiology ( Site 0002), New York, New York
  - Lillestol Research ( Site 0026), Fargo, North Dakota
  - altoona center for clinical research ( Site 0089), Duncansville, Pennsylvania
  - Cardiology Consultants of Philadelphia Yardley ( Site 0097), Yardley, Pennsylvania
  - Piedmont Research Partners ( Site 0090), Fort Mill, South Carolina
  - Velocity Clinical Research, Greenville ( Site 0023), Greenville, South Carolina
  - Coastal Carolina Research Center ( Site 0006), North Charleston, South Carolina
  - Monument Health Clinical Research, a department of Monument -Monument Health Clinical Research, a d ( Site 0009), Rapid City, South Dakota
  - Holston Medical Group ( Site 0048), Kingsport, Tennessee
  - Alliance for Multispecialty Research, LLC ( Site 0008), Knoxville, Tennessee
  - Velocity Clinical Research, Dallas ( Site 0114), Dallas, Texas
  - Center for Cardiometabolic Disease Prevention/Baylor College of Medicine ( Site 0111), Houston, Texas
  - Clinical Trials of Texas, LLC ( Site 0103), San Antonio, Texas
  - Synexus Clinical Research US, Inc. ( Site 0110), Salt Lake City, Utah
  - Velocity Clinical Research, Salt Lake City ( Site 0019), West Jordan, Utah
  - Manassas Clinical Research Center ( Site 0007), Manassas, Virginia
  - Health Research of Hampton Roads, Inc. ( Site 0044), Newport News, Virginia
  - Alliance for Multispecialty Research, LLC ( Site 0101), Norfolk, Virginia
  - National Clinical Research, Inc ( Site 0061), Richmond, Virginia
  - Centricity Research Suffolk Family Medicine ( Site 0092), Suffolk, Virginia
  - Rainier Clinical Research Center ( Site 0116), Renton, Washington
- Argentina (6):
  - CEDIC ( Site 0612), CABA, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0605), Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate ( Site 0600), Zárate, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada ( Site 0604), Buenos Aires, Buenos Aires F.D.
  - Fundación Respirar ( Site 0610), Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Metabólicas (CINME)-Cardiology ( Site 0620), CABA
- China (18):
  - Beijing Anzhen Hospital, Capital Medical University-Cardiovascular ( Site 3300), Beijing, Beijing Municipality
  - Beijing Friendship Hospital Affiliate of Capital University-Cardiology ( Site 3303), Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University ( Site 3320), Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital ( Site 3321), Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital-Cardiology ( Site 3304), Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University ( Site 3329), Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital ( Site 3379), Huizhou, Guangdong
  - The University of Hong Kong-Shenzhen Hospital-Cardiovascular department ( Site 3318), Shenzhen, Guangdong
  - Jingzhou Central Hospital-Cardiology ( Site 3376), Jingzhou, Hubei
  - Wuhan Fourth Hospital ( Site 3356), Wuhan, Hubei
  - Hunan Provincial People's Hospital-Cardiology ( Site 3317), Changsha, Hunan
  - Changzhou Second People's Hospital-Cardiology ( Site 3373), Changzhou, Jiangsu
  - Northern Jiangsu People's Hospital ( Site 3308), Yangzhou, Jiangsu
  - The Third Hospital of Nanchang - Fuhe-cardiology ( Site 3378), Nanchang, Jiangxi
  - Siping Central People's Hospital-Cardiovascular Department ( Site 3311), Siping, Jilin
  - Xianyang Hospital of Yan'an University ( Site 3340), Xianyang, Shaanxi
  - Chengdu Second Municipal People's Hospital ( Site 3332), Chengdu, Sichuan
  - People's Hospital of Lishui City-department of cardiovascular ( Site 3302), Lishui, Zhejiang
- Colombia (6):
  - Fundación Centro de Investigación Clínica CIC ( Site 0906), Medellín, Antioquia
  - Ciensalud Ips S A S ( Site 0903), Barranquilla, Atlántico
  - Clinica de la Costa S.A.S. ( Site 0902), Barranquilla, Atlántico
  - Salud SURA Calle 100 ( Site 0918), Bogotá, Cundinamarca
  - Healthy Medical Center S.A.S ( Site 0913), Zipaquirá, Cundinamarca
  - Fundación Valle del Lili ( Site 0904), Cali, Valle del Cauca Department
- Germany (6):
  - Unterfrintroper Hausarztzentrum Klinische Forschung ( Site 1542), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Universitätsstudienzentrum für Stoffwechselerkranku ( Site 1508), Dresden, Saxony
  - Hausarzt- und Diabetologische Schwerpunktpraxis Hohenmölsen - Weiβenfels ( Site 1527), Hohenmölsen, Saxony-Anhalt
  - Zentralklinik Bad Berka ( Site 1530), Bad Berka, Thuringia
  - Velocity Clinical Research GmbH Berlin ( Site 1502), Berlin
  - Charite Universitätsmedizin Berlin Campus Benjamin Franklin ( Site 1533), Berlin
- Israel (9):
  - Hillel Yaffe Medical Center ( Site 1705), Hadera
  - Rambam Health Care Campus-internal department ( Site 1718), Haifa
  - Shaare Zedek Medical Center ( Site 1710), Jerusalem
  - Hadassah Medical Center ( Site 1706), Jerusalem
  - Hadassah Medical Center ( Site 1709), Jerusalem
  - Meir Medical Center. ( Site 1714), Kfar Saba
  - Rabin Medical Center ( Site 1720), Petah Tikva
  - Sheba Medical Center ( Site 1708), Ramat Gan
  - Yitzhak Shamir Medical Center. ( Site 1712), Ẕerifin
- Italy (6):
  - Fondazione Policlinico Tor Vergata ( Site 1809), Rome, Lazio
  - Centro Cardiologico Monzino ( Site 1804), Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda-Unità Ricerche Cliniche della Cardiologia 4 ( Site 1811), Milan, Milano
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino ( Site 1801), Turin, Piedmont
  - Azienda Ospedaliera Sant'Andrea-Department of Clinical and Molecular Medicine ( Site 1807), Rome, Roma
  - Azienda Ospedaliera Garibaldi ( Site 1810), Catania
- Japan (23):
  - Hirohata Naika Clinic ( Site 3513), Kitakyusyu-shi, Fukuoka
  - Nakakinen clinic ( Site 3510), Naka, Ibaraki
  - Noritake Clinic ( Site 3512), Ushiku, Ibaraki
  - National Hospital Organization Kanazawa Medical Center ( Site 3508), Kanazawa, Ishikawa-ken
  - Hirano Medical Clinic ( Site 3522), Morioka, Iwate
  - Shirai Healthcare Clinic Izumichuou ( Site 3527), Sendai, Miyagi
  - Rinku General Medical Center ( Site 3503), Izumisano, Osaka
  - Shiraiwa Medical Clinic ( Site 3514), Kashihara, Osaka
  - Medical Corporation Heishinkai OCROM Clinic ( Site 3501), Suita-shi, Osaka
  - Saitama Medical University Hospital ( Site 3506), Iruma, Saitama
  - Teramoto Medical and Dental Clinic ( Site 3507), Bunkyo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic ( Site 3505), Chuo-ku, Tokyo
  - Fukuwa Clinic ( Site 3504), Chuo-ku, Tokyo
  - Teikyo University Hospital ( Site 3500), Itabashi-ku, Tokyo
  - Kato Clinic of Internal Medicine ( Site 3509), Katsushika-ku, Tokyo
  - Kanno Naika ( Site 3511), Mitaka, Tokyo
  - Sugawara Clinic ( Site 3519), Nerima-ku, Tokyo
  - Shin Clinic ( Site 3517), Ōta-ku, Tokyo
  - Medical Corporation Heishinkai ToCROM Clinic ( Site 3502), Shinjuku-ku, Tokyo
  - Mitsukoshi Health and Welfare Foundation ( Site 3521), Shinjuku-ku, Tokyo
  - Medical Corporation Hakuaikai Wellness Tenjin Clinic ( Site 3520), Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital ( Site 3518), Hiroshima
  - Mishuku Hospital ( Site 3524), Tokyo
- Mexico (2):
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad-Endocrinology ( Site 1057), Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 1071), Mexico City, Mexico City
- South Africa (6):
  - IATROS INTERNATIONAL ( Site 2247), Bloemfontein, Free State
  - Soweto Clinical Trials Centre ( Site 2242), Johannesburg, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital-WCR-LIPIDS ( Site 2241), Johannesburg, Gauteng
  - Tiervlei Trial Centre-Clinical ( Site 2246), Bellville, Cape Town, Western Cape
  - TREAD Research ( Site 2253), Cape Town, Western Cape
  - University of Cape Town (UCT)-Medicine, Division of Lipidology ( Site 2259), Cape Town, Western Cape
- South Korea (15):
  - Wonju Severance Christian Hospital ( Site 3008), Wŏnju, Kang-won-do
  - Chonnam National University Hospital ( Site 3014), Gwangju, Kwangju-Kwangyokshi
  - Seoul National University Bundang Hospital ( Site 3005), Seongnam, Kyonggi-do
  - Ajou University Hospital ( Site 3006), Suwon, Kyonggi-do
  - Chungbuk National University Hospital ( Site 3011), Cheongju-si, North Chungcheong
  - Dong-A University Hospital ( Site 3013), Busan, Pusan-Kwangyokshi
  - Pusan National University Hospital-Internal Medicine ( Site 3012), Busan, Pusan-Kwangyokshi
  - Inje University Haeundae Paik Hospital ( Site 3010), Haeundae-gu, Pusan-Kwangyokshi
  - Keimyung University Dongsan Hospital CRC room 1 ( Site 3003), Daegu, Taegu-Kwangyokshi
  - Seoul National University Hospital ( Site 3001), Seoul
  - Kangbuk Samsung Hospital ( Site 3009), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 3002), Seoul
  - Asan Medical Center ( Site 3004), Seoul
  - Samsung Medical Center-cardiology ( Site 3000), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital-cardiology ( Site 3007), Seoul
- Spain (9):
  - Hospital Universitario Virgen Macarena ( Site 2352), Seville, Andalusia
  - EBA CENTELLES ( Site 2311), Centelles, Catalonia
  - Hospital Abente y Lago ( Site 2356), A Coruña, La Coruna
  - CHUS - Hospital Clinico Universitario-Cardiology - Clinical Research Unit ( Site 2320), Santiago de Compostela, La Coruna
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-Endocrinologia y Nutrición ( Site 2344), Pozuelo de Alarcón, Madrid
  - Hospital Universitario Fundacion ALcorcon-Endocrinologia y Nutrición ( Site 2316), Alcorcón, Madrid, Comunidad de
  - Vithas Hospital Sevilla-Unidad de Salud Metabólica. Diabetes y Obesidad ( Site 2349), Castilleja de la Cuesta, Sevilla
  - HOSPITAL CLINICO DE VALENCIA-CARDIOLOGY ( Site 2321), Valencia, Valenciana, Comunitat
  - Hospital Universitario 12 de Octubre-Internal Medicine. Unidad de Ensayos Clínicos ( Site 2319), Madrid
- Taiwan (7):
  - Chi Mei Medical Center-Cardiology ( Site 3104), Tainan, Tainan
  - Changhua Christian Hospital ( Site 3101), Changhua
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 3102), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 3107), Tainan
  - National Taiwan University Hospital ( Site 3100), Taipei
  - Taipei Medical University Hospital-Cardiology ( Site 3108), Taipei
  - Taipei Veterans General Hospital ( Site 3106), Taipei
- Turkey (Türkiye) (6):
  - Hacettepe Universite Hastaneleri ( Site 2500), Altindağ, Ankara
  - Ege Universitesi Hastanesi-Cardilogy Department ( Site 2502), Bornova, İzmir
  - Ankara Bilkent Şehir Hastanesi-cardiology ( Site 2501), Ankara
  - Eskisehir Osmangazi University-Cardiology ( Site 2510), Eskişehir
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri-endocrine ( Site 2522), Kayseri
  - Kocaeli Üniversitesi-Cardiology ( Site 2516), Kocaeli

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26172&tenant=MT_MSD_9011